CLINICAL TRIAL: NCT04912271
Title: Granisetron Transdermal Delivery System Versus Palonosetron in the Prevention of Delayed Chemotherapy-induced Nausea and Vomiting: a Phase 3 Non-inferiority Randomized Trial
Brief Title: Granisetron Transdermal Patch for Prophylaxis of Delayed CINV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YBCSG-21-04
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Chemotherapy-induced Nausea and Vomiting (CINV)
Keywords: delayed CINV; granisetron transdermal delivery system
MeSH Terms: conditions — Vomiting | interventions — Granisetron; Palonosetron; Aprepitant; fosaprepitant; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granisetron transdermal patch (other name: sancuso), aprepitant or fosaprepitant, dexamethasone (Experimental): Patients received granisetron transdermal patch plus dexamethasone followed by oral aprepitant or fosaprepitant infusion Granisetron transdermal patch Aprepitant 125 mg PO D1, 80 mg PO D2-D3; Fosaprepitant 150 mg IV D1 Dexamethasone 7.5-10 mg IV/PO D1
  Interventions: Drug: Granisetron transdermal patch; Drug: Aprepitant; Drug: Fosaprepitant; Drug: Dexamethasone
- Palonosetron, aprepitant or fosaprepitant, dexamethasone (Active Comparator): Patients received intravenous palonosetron plus dexamethasone followed by oral aprepitant or fosaprepitant infusion Palonosetron 0.25 mg IV D1 Aprepitant 125 mg PO D1, 80 mg PO D2-D3; Fosaprepitant 150 mg IV D1 Dexamethasone 7.5-10 mg IV/PO D1
  Interventions: Drug: Palonosetron; Drug: Aprepitant; Drug: Fosaprepitant; Drug: Dexamethasone

INTERVENTIONS:
Drug: Granisetron transdermal patch — Granisetron transdermal delivery system (GTDS) is the first 5-HT3 drug to be transdermally delivered and represents a convenient alternative to oral and intravenous antiemetics for the treatment of chemotherapy-induced nausea and vomiting.
  Other Names: sancuso
  Arms: Granisetron transdermal patch (other name: sancuso), aprepitant or fosaprepitant, dexamethasone
Drug: Palonosetron — Palonosetron is a second-generation 5-HT3 receptor antagonist with proposed higher efficacy and sustained action for prophylaxis of postoperative nausea and vomiting (PONV).
  Arms: Palonosetron, aprepitant or fosaprepitant, dexamethasone
Drug: Aprepitant — Aprepitant is a licensed treatment for nausea and vomiting, which blocks substance P activation of NK-1 (neurokinin 1) receptors.
Drug: Fosaprepitant — Fosaprepitant is a neurokinin-1 receptor antagonist, approved for the prevention of chemotherapy-induced nausea and vomiting.
Drug: Dexamethasone — Dexamethasone, one of the glucocorticoids, has been suggested as a first-line drug for preventing low-level emetogenic chemotherapy- and radiotherapy-induced nausea and vomiting.

SUMMARY:
Transdermal granisetron has been shown to as effective as oral/ intravenous granisetron when administered with or without dexamethasone. However, it has not been evaluated specifically against the delayed response of chemotherapy-induced nausea and vomiting (CINV) in comparison with palonosetron, as the complete response for the delayed phase was not reported in the comparative study by Seol et al (Support Care Cancer 2016;24:945-952). Thus, transdermal granisetron needs to be compared with palonosetron as part of dual and triple therapy in the delayed phase of CINV.

This investigator-initiated study aims to compare the efficacy of granisetron transdermal patch and palonosetron combined with NK-1 receptor antagonist and dexamethasone in the prevention of delayed CINV in Chinese breast cancer patients who received high emetic or moderate emetic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥ 18 years;
2. Pathologically confirmed breast cancer;
3. The physical status score ECOG ≤ 2;
4. Life expectancy of ≥3 months;
5. Patients first or had already received chemotherapy;
6. Patients scheduled to receive HEC/MEC chemotherapy, and the main emetic drugs will be used within a single day;
7. Patients first use of granisetron transdermal patch;
8. In accordance with the indication of chemotherapy and basic requirements;

   * Peripheral haematology: Hb ≥8.0g/dL; absolute neutrophil count≥1.5×109/L; platelet count ≥80×109/L
   * Blood biochemistry: Total bilirubin < 1.5×ULN, ALT and AST ≤ 2.5×ULN; if liver metastasis, ALT and AST < 5×ULN, creatinine ≤ 1.5×ULN
9. Patients voluntarily participate and sign the informed consent form;
10. Be able to read, understand and complete patient diaries independently.

Exclusion Criteria:

1. Contraindicated to 5-HT receptor antagonists, NK-1 receptor antagonist or dexamethasone;
2. Patients have used 5-HT receptor antagonist, NK1 receptor antagonist or any study drugs within 4 weeks before chemotherapy
3. Any nausea and vomiting (II or above) within 72 hours before the start of chemotherapy;
4. According to the judgment of the investigators, there are concomitant diseases (including but not limited to hypertension, severe diabetes, active infection, thyroid disease, etc.) that seriously endanger the safety of the patient or affect the completion of the study;
5. Patients scheduled to receive radiotherapy of whole body, brain or upper abdomen;
6. Confirmed by craniocerebral CT or MRI, patients with brain tumor lesions or patients taking drugs to treat brain tumors or epileptic symptoms;
7. History of drug abuse and alcohol dependence;
8. Pregnancy, lactation or intended pregnancy;
9. History of allergic reactions to drugs with similar chemical structures, or to transdermal therapeutic systems, including commercial dressings such as Elastoplast®
10. Unable to swallow, having intestinal obstruction, or other factors that affect the taking and absorption of the drug;
11. Long-term use of any inhibitors or inducers of CYP3A4, or take these drugs within 4 weeks before the first day of chemotherapy;
12. Other situations evaluated by investigators as unsuitable for enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2021-06-10 (Estimated); Primary Completion 2022-06-10 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) in delay phase of CINV | From 24 hours after initiating administration of chemotherapy agents to day 7 (24-168 hours)
  To compare the complete response (CR) of Granisetron transdermal patch to Palonosetron (complete response is defined as no vomiting and no rescue medication) in delay phase of CINV

SECONDARY OUTCOMES:
complete response (CR) in the acute and overall phase of CINV | From 24 hours after initiating administration of chemotherapy agents to day 7 (24-168 hours)
  1. To compare the complete response (CR) of Granisetron transdermal patch to Palonosetron (complete response is defined as no vomiting and no rescue medication) in the acute and overall phase of CINV
complete control (CC) in delay phase of CINV | From 24 hours after initiating administration of chemotherapy agents to day 7 (24-168 hours)
  2. To compare the complete control (CC) of Granisetron transdermal patch to Palonosetron (complete control is defined as no vomiting, mild nausea and no rescue medication) in delay phase of CINV
complete control (CC) in the acute and overall phase of CINV | From initiating administration of chemotherapy agents to day 1 (0-24 hours) and day 7 (0-168 hours)
  3. To compare the complete control (CC) of Granisetron transdermal patch to Palonosetron (complete control is defined as no vomiting and no rescue medication) in the acute and overall phase of CINV
Patients' satisfaction with antiemetic therapy (assessed using a 10-cm visual analog scale at the time of patch removal | 7 days
  "dissatisfied" on the left end (0 cm) of visual analog scale and the "very satisfied" on the right end of visual analog scale (10 cm)

REFERENCES:
- [Derived] Liu X, Meng Y, Du Y, Mu Y, Li G, Li H, Guan X, Zhang J. Granisetron transdermal delivery system versus palonosetron in the prevention of long-delayed nausea and vomiting: a phase III randomized trial. Oncologist. 2026 Feb 5;31(3):oyag007. doi: 10.1093/oncolo/oyag007. PMID 41520166